CLINICAL TRIAL: NCT06639971
Title: Retrospective Cohort Study on the Therapeutic Effects of Immunotherapy and Targeted Therapy Combined With or Without Radiotherapy for Hepatocellular Carcinoma Based on Real-world Data
Brief Title: Therapeutic Effects of Immuno-targeted Therapy Combined With or Without RT for HCC
Acronym: RIO-HCC
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2024447; B2024-336R (Other: Zhongshan Hospital, Fudan University)
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular Carcinoma; Radiotherapy; Immunotherapy; Target therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ITR group: hepatocellular carcinoma patients treated with immunotherapy and targeted therapy combined with radiotherapy
- IT group: hepatocellular carcinoma patients treated with immunotherapy and targeted therapy alone

SUMMARY:
The objective of this retrospective cohort study is to investigate the therapeutic effects of combined immunotherapy and targeted therapy, with or without radiotherapy, in patients with hepatocellular carcinoma.

The main question it aims to answer is:

Does the addition of radiotherapy to immunotherapy and targeted therapy enhance the therapeutic effect more significantly compared to immunotherapy and targeted therapy alone for patients with hepatocellular carcinoma?

DETAILED DESCRIPTION:
A retrospective analysis will be conducted on the clinical data of patients with hepatocellular carcinoma who underwent combined immunotherapy and targeted therapy with radiotherapy, as well as those who received immunotherapy and targeted therapy alone, at Zhongshan Hospital, Fudan University, from January 1, 2017, to December 31, 2023. The pmary objective is to assess the disparities in treatment efficacy and treatment-related adverse events between the two cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatocellular carcinoma confirmed by histopathological/cytopathological examination, or fulfilling the clinical diagnostic criteria for primary liver cancer according to the Guidelines for Diagnosis and Treatment of Primary Liver Cancer (2024 edition).
2. Patients with hepatocellular carcinoma who received targeted therapy and immunotherapy at Zhongshan Hospital affiliated with Fudan University from January 1, 2017, to December 31, 2023.
3. Tumor staging meeting at least one of the following criteria: 1) CNLC stage IIIa or IIIb hepatocellular carcinoma with concurrent vascular invasion or extrahepatic metastasis; 2) CNLC stage IIb hepatocellular carcinoma presenting as a localized lesion unsuitable for surgical resection or transarterial chemoembolization (TACE); 3) Presence of main portal vein or inferior vena cava tumor thrombus; 4) Disease progression observed after multiple local treatments (such as surgical resection, TACE, radiofrequency ablation, etc.).
4. Availability of complete clinical and follow-up information.
5. Patients have provided informed consent for donation of biological samples, allowing the donated samples and related information to be used for all medical research purposes.

Exclusion Criteria:

1. Contraindications for radiotherapy include hepatocellular carcinoma with diffuse intrahepatic lesions, PS score of 3-4, Child-Pugh C liver function, or the presence of severe underlying medical conditions.
2. Known components of the patient population include cholangiocarcinoma (ICC), mixed hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, or fibrolamellar carcinoma.
3. Exclusion criteria encompass a history of malignancies other than hepatocellular carcinoma within the past 5 years, except for limited-stage tumors considered cured, such as cervical carcinoma in situ, basal cell carcinoma, and prostate carcinoma in situ.
4. Any other circumstances that the investigator deems unsuitable for participation in the study are also exclusion criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes HCC patients who received targeted therapy and immunotherapy at Zhongshan Hospital affiliated with Fudan University between January 1, 2017, and December 31, 2023. Tumor staging criteria included CNLC stage IIIa or IIIb hepatocellular carcinoma with concurrent vascular invasion or extrahepatic metastasis, CNLC stage IIb hepatocellular carcinoma presenting as a localized lesion unsuitable for surgical resection or transarterial chemoembolization (TACE), presence of main portal vein or inferior vena cava tumor thrombus, or disease progression after multiple local treatments.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Up to 2 years
  Progression free survival is defined as the duration between the date of of initial administration of targeted therapy and immunotherapy to the date of first documented progression or death due to any cause or date of last follow-up, whichever is earlier.

SECONDARY OUTCOMES:
Overall Survival | Up to 2 years
  Overall survival is defined as the duration between the date of initial administration of targeted therapy and immunotherapy to the date of death due to any cause or the date of last follow-up, whichever is earlier.
Treatment-related Adverse Effects | Up to 2 years
  At baseline and at subsequent follow up till 2 years based on Common Terminology Criteria for Adverse Events 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with other researchers in order to protect patients' privacy.

REFERENCES:
- [Background] Zhong L, Wu D, Peng W, Sheng H, Xiao Y, Zhang X, Wang Y. Safety of PD-1/PD-L1 Inhibitors Combined With Palliative Radiotherapy and Anti-Angiogenic Therapy in Advanced Hepatocellular Carcinoma. Front Oncol. 2021 May 19;11:686621. doi: 10.3389/fonc.2021.686621. eCollection 2021. PMID 34094988
- [Background] Su K, Guo L, Ma W, Wang J, Xie Y, Rao M, Zhang J, Li X, Wen L, Li B, Yang X, Song Y, Huang W, Chi H, Gu T, Xu K, Liu Y, Chen J, Wu Z, Jiang Y, Li H, Zeng H, Wang P, Feng X, Chen S, Yang B, Jin H, He K, Han Y. PD-1 inhibitors plus anti-angiogenic therapy with or without intensity-modulated radiotherapy for advanced hepatocellular carcinoma: A propensity score matching study. Front Immunol. 2022 Sep 23;13:972503. doi: 10.3389/fimmu.2022.972503. eCollection 2022. PMID 36211350
- [Background] Ren Z, Xu J, Bai Y, Xu A, Cang S, Du C, Li Q, Lu Y, Chen Y, Guo Y, Chen Z, Liu B, Jia W, Wu J, Wang J, Shao G, Zhang B, Shan Y, Meng Z, Wu J, Gu S, Yang W, Liu C, Shi X, Gao Z, Yin T, Cui J, Huang M, Xing B, Mao Y, Teng G, Qin Y, Wang J, Xia F, Yin G, Yang Y, Chen M, Wang Y, Zhou H, Fan J; ORIENT-32 study group. Sintilimab plus a bevacizumab biosimilar (IBI305) versus sorafenib in unresectable hepatocellular carcinoma (ORIENT-32): a randomised, open-label, phase 2-3 study. Lancet Oncol. 2021 Jul;22(7):977-990. doi: 10.1016/S1470-2045(21)00252-7. Epub 2021 Jun 15. PMID 34143971